CLINICAL TRIAL: NCT05682365
Title: Effectiveness of an Online Personalized Intervention Based on a Risk Algorithm for the Universal Prevention of Anxiety: Randomized Controlled Trial. The prevANS Study.
Brief Title: Online Personalized Intervention for the Prevention of Anxiety.
Acronym: prevANS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Collaborators: Agencia Estatal de Investigación (AEI) (Unknown); Institute of Health Carlos III (ISCIII) (Unknown); Institute of Biomedical Research in Málaga (IBIMA) (Unknown); European Regional Development Fund (Other)
Responsible Party: Principal Investigator, Patricia Moreno Peral, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PID2020-119652RA-I00
Record Dates: First submitted 2022-12-08; First posted 2023-01-12 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Disorders
Keywords: Anxiety Disorders; Primary prevention; Randomized controlled trial; m-Health; e-Health
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prevANS intervention (Experimental): In this arm, participants will receive an online personalized intervention to prevent anxiety disorders based on a risk predictive algorithm (predictA).
  Interventions: Behavioral: prevANS intervention
- Control group (No Intervention): In this arm, participants will continue receiving the usual care from their health providers. However, they will not receive any intervention, but they will fill out the same questionnaires as in the intervention group.

INTERVENTIONS:
Behavioral: prevANS intervention — prevANS intervention will be self-guided and can be implemented from the prevANS web or from the participants' Smartphone (through an APP). The prevANS intervention will have different intensities depending on the risk level of the population, evaluated from the already validated risk algorithm for anxiety: predictA. Participants will be classified as moderate-high or low risk of anxiety. Both groups of risk will receive information on their level and profile (risk factors) of anxiety and psychoeducational information periodically; also, they will work towards manage stressors and enhance protective factors. However, participants with moderate-high risk of anxiety will also receive a cognitive-behavioral training (problem solving, decision-making, handling thoughts / concerns and emotions and communicational skills).
  Arms: prevANS intervention

SUMMARY:
Objective: To design, develop and evaluate an online personalized intervention based on a risk algorithm for the universal prevention of anxiety disorders in the general population.

Methods: Randomized controlled trial, with two parallel arms and 12 months follow-up. The entire process of recruitment, randomization, intervention and follow-up will be carried out from a web platform designed for the study (web prevANS). Through a communication campaign, where announcements and informative videos will be produced, and through the dissemination on prevANS website, 2,000 Spanish and Portuguese adult participants without anxiety in the baseline of the study will be recruited. The participants will be randomly assigned to the prevANS intervention, which will be self-guided and can be implemented from the prevANS web or from the participants' Smartphone (through an APP), or to a control group. The prevANS intervention will have different intensities depending on the risk level of the population, evaluated from the already validated risk algorithm for anxiety: predictA. Participants with a low risk of anxiety will receive information on their level and profile (risk factors) of anxiety and psychoeducational information periodically. Participants with moderate and high risk of anxiety will also receive information on their risk level and profile, but will also include a cognitive-behavioral training (problem solving, decision-making, handling thoughts / concerns and emotions and communicational skills). Both groups of risk will work towards manage stressors and enhance protective factors. The control group will not receive any intervention, but they will fill out the same questionnaires as in the intervention group. The main result will be the incidence of new cases of anxiety disorders measured by CIDI, and the secondary results will be the reduction of anxiety (GAD-7) and depression (PHQ-9) symptoms, of the risk probability of anxiety and depression (predictA and predictD algorithms) and improvement of quality of life measured by SF-12 and EuroQol, and cost-effectiveness and cost-utility.

ELIGIBILITY:
Inclusion Criteria:

* GAD-7 <10 at baseline
* GAD-7 ≥10 at baseline and a negative diagnosis of anxiety disorders by CIDI

Exclusion Criteria:

* Not have a smartphone and internet for personal use
* Unable to speak Spanish
* Documented terminal illness
* Documented cognitive impairment
* Documented serious mental illness (psychosis, bipolar, addictions, etc.)
* Being involved in any psychological intervention or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 12 months
  Rate of anxiety disorders measured by the Composite International Diagnostic Interview (CIDI). CIDI is a structured diagnostic interview that provides current diagnoses of anxiety disorders according to DSM.

SECONDARY OUTCOMES:
Anxious symptoms measured by the General Anxiety Questionnaire (GAD-7) | 12 months
  The General Anxiety Questionnaire (GAD-7) measures generalized anxiety disorder through 7 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of anxiety, the scale range is 0 to 21 (7 items).
Depressive symptoms measured by the Patient Health Questionnaire-9 (PHQ-9) | 12 months
  The Patient Health Questionnaire-9 (PHQ-9) measures symptoms of depression through 9 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of depression, the scalen range is 0 to 27 (9 items).
Probability of anxiety measured by the Spanish predictA risk algorithm | 12 months
  The Spanish predictA risk algorithm measures 12 risk factors for anxiety disorders
Probability of depression measured by the Spanish predictD risk algorithm | 12 months
  The Spanish predictD risk algorithm measures 13 risk factors for depression
Quality of life measured by SF-12 | 12 months
  The 12-item Short Form (SF-12) measures quality of life related to physical health and quality of life related to mental health. Scores on the scales range from 0 to 100. Higher scores are equivalent to better health-related quality of life.
Cost-effectiveness | 12 months
  It will be conducted from two perspectives: (1) a societal perspective and (2) a National Health System perspective. We will calculate incremental cost-effectiveness ratio (ICER) using the incremental cost (difference in costs between arms) divided by incremental effectiveness (difference in the number of diagnoses of anxiety disorders between arms).
Cost-utility | 12 months
  It will be conducted from two perspectives: (1) a societal perspective and (2) a National Health System perspective. We will calculate incremental cost-effectiveness ratio (ICER) using the incremental cost (difference in costs between arms) divided by incremental QALYs (difference in QALYs between arms). Quality-adjusted life years (QALYs) will be measured using the EuroQol five questionnaire (EuroQol-5D).
Acceptability and satisfaction with the intervention (prevANS intervention) measured by u-MARS scale | 12 months
  The User Version of the Mobile Application Rating Scale (u-MARS) consists of 23 items assessing app quality, each of which is scored 1 ('poor') to 5('excellent'), except items 14-17 and item 19, which also include the "not applicable" option. Higher scores are equivalent to higher app quality.
Mediator of the intervention: cognitive change | 12 months
  The cognitive change will be evaluated through the number of negative thoughts worked and modified in the app
Subgroup analysis according to age | 12 months
  A subgroup analysis will be conducted according to age of the participants (from 18 to 30 years; from 31 to 50 years; and > 50 years)
Subgroup analysis according to sex | 12 months
  A subgroup analysis will be conducted according to sex of the participants (women or men)
Subgroup analysis according to education level | 12 months
  A subgroup analysis will be conducted according to education level of the participants (without primary education; primary education; secondary education; or higher education)
Subgroup analysis according to anxiety symptoms at baseline (through the GAD-7 questionnaire) | 12 months
  The General Anxiety Questionnaire (GAD-7) measures generalized anxiety disorder through 7 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of anxiety, the scale range is 0 to 21 (7 items). The subgroups will be: 1) from 0 to 5 points; and 2) > 5 points
Subgroup analysis according to depressive symptoms at baseline (through the PHQ-9 questionnaire) | 12 months
  The Patient Health Questionnaire-9 (PHQ-9) measures symptoms of depression through 9 items, each of which is scored 0 ('not at all') to 3 ('nearly every day'). Low scores are equivalent to less symptoms of depression, the scalen range is 0 to 27 (9 items). The subgroups will be: 1) from 0 to 5 points; 2) from 6 to 10 points; and 3) > 10 points
Subgroup analysis according to risk level of anxiety (through the predictA risk algorithm) | 12 months
  The Spanish predictA risk algorithm measures 12 risk factors for anxiety disorders. The subgroups will be: 1) probability of risk from 0 to 6%; and 2) probability of risk >6%
Subgroup analysis according to risk level of depression (through the predictD risk algorithm) | 12 months
  The Spanish predictD risk algorithm measures 13 risk factors for depression. The subgroups will be: 1) probability of risk from 0 to 9%; and 2) probability of risk >9%

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Moreno-Peral, PhD, Principal Investigator — University of Malaga
Locations (1):
- Facultad de Psicología y Logopedia, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data generated during this study will include detailed information on the protocols and analyses used to allow their reproducibility and future analyses by other groups. The data generated from this research will be made available to affiliated investigators through secure and anonymized databases. Only investigators with specific independent ethics committee approval will have access to any anonymized data. The research coordinator of the prevANS study can be contacted for de-identified data requests. Consent for such data sharing will be integral to enrollment in the study, and our participants will be asked about their willingness to have their data shared to advance health research.

REFERENCES:
- [Derived] Moreno-Peral P, Rodriguez-Morejon A, Bellon JA, Garcia-Huercano C, Martinez-Vispo C, Campos-Paino H, Galan S, Reyes-Martin S, Sanchez Aguadero N, Rangel-Henriques M, Motrico E, Conejo-Ceron S. Effectiveness of a universal personalized intervention for the prevention of anxiety disorders: Protocol of a randomized controlled trial (the prevANS project). Internet Interv. 2023 Jun 22;34:100640. doi: 10.1016/j.invent.2023.100640. eCollection 2023 Dec. PMID 38023964